CLINICAL TRIAL: NCT01157195
Title: Home-Based Automated Therapy of Arm Function After Stroke Via Tele-Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gitendra Uswatte, Associate Professor of Psychology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F071227003; R01HD053750 (NIH)
Record Dates: First submitted 2010-06-17; First posted 2010-07-05 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: stroke; chronic; arm; rehabilitation; tele-health
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CI therapy (Active Comparator)
  Interventions: Behavioral: CI therapy
- Tele-AutoCITE (Experimental): AutoCITE stands for Automated Constraint Induced Therapy Extender.
  Interventions: Behavioral: Tele-AutoCITE

INTERVENTIONS:
Behavioral: Tele-AutoCITE — Automated, remotely-administered form of CI therapy
  Arms: Tele-AutoCITE
Behavioral: CI therapy — CI therapy is a behavioral approach to physical rehabilitation that has three components: 1. intense training of the more affected arm for several hours daily for multiple consecutive days, 2. restraint of the less affected arm during training hours and afterwards during the treatment period, 3. A package of behavioral techniques designed to transfer gains from the treatment setting to daily life. In this trial, CI therapy will be administered for 3 1/2 hours per day for 10 consecutive weekdays.
  Arms: CI therapy

SUMMARY:
Constraint-Induced Movement therapy, also known as CI therapy, is an approach to physical rehabilitation derived from basic behavioral and neuroscience research. It has been shown to be efficacious for rehabilitating use of the more-affected arm in individuals more than one year after stroke with mild to moderate motor impairment. The first component of the therapy is intensive training in use of the more-affected arm on functional tasks for 3 hours daily for 10 consecutive weekdays. The second is wearing a protective safety mitt on the less-affected hand for all waking hours of the approximately 2-week treatment period that it is safe to do so. The purpose of the mitt is to discourage use of the less-affected arm. The third is a group of behavioral techniques designed to transfer gains from the treatment setting to the real world, which takes a therapist, on average, 30 minutes to implement on each treatment day.

The purpose of this project is to develop and test a method for automating the delivery of this efficacious treatment in a way that the therapy can be provided in stroke patients' homes. After developing an automated CI therapy workstation that has tele-health capabilities, the investigators will conduct a randomized controlled trial to evaluate whether CI therapy delivered in the home using this workstation with remote supervision by a therapist via an Internet-based audiovisual link provides outcomes that are just as good as CI therapy delivered by a "live" therapist.

ELIGIBILITY:
Inclusion Criteria:

* more than 1 year after stroke
* some ability to voluntarily open fingers on more affected side of body
* some ability to voluntarily raise wrist on more affected side of body
* ability to stand independently for two minutes
* ability to transfer from sit to stand independently

Exclusion Criteria:

* serious, concurrent medical conditions including frailty
* excessive spasticity (high muscle tone) in more affected arm
* impairment in thinking that makes compliance with study activities difficult

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Motor Activity Log (MAL) Arm Use Scale at 2 weeks | Baseline to 2 weeks (average)
  Well-validated structured interview that assesses how much and how well the more-affected arm after stroke has been used to accomplish everyday activities over a specified period.

SECONDARY OUTCOMES:
Change in Wolf Motor Function Test (WMFT) Performance Rate at 2 weeks | Baseline to 2 weeks (average)
  Well-validated laboratory motor performance test that assesses how quickly an individual can perform upper-extremity tasks with the more-affected arm after stroke.
Change in MAL Arm Use Scale at 6 months | Baseline to 6 months (average)
  See primary outcome.
Change in MAL Arm Use Scale at 12 months | Baseline to 12 months (average)
  See primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gitendra Uswatte, PhD, Principal Investigator — Psychology Department, University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Taub E, Uswatte G, Pidikiti R. Constraint-Induced Movement Therapy: a new family of techniques with broad application to physical rehabilitation--a clinical review. J Rehabil Res Dev. 1999 Jul;36(3):237-51. PMID 10659807